CLINICAL TRIAL: NCT07226310
Title: The Hysterosalpingogram (HSG) Experience And Tubal Spasm (HEAT) Study: A Randomized Controlled Trial
Brief Title: The Hysterosalpingogram (HSG) Experience And Tubal Spasm (HEAT) Study
Acronym: HEAT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18943
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to warmed vs cold (room temperature) HSG,
Who Masked: Participant, Investigator
Masking Description: This study will be blinded in a manner that the research nurse, patient, and provider will not be aware of patient allocation at time of recruitment and enrollment. The patient will be assigned a unique study ID number and the randomization module in REDCap will be used to assign the participant to either the experimental (warm) or control (cold) group.
  The patient will remain blinded to the treatment allocation but the research nurse and performing provider will be unblinded to allow for correct choice and use of warm versus cold contrast media. As both the research nurse and provider will touch the HSG contrast media and be able to discern if it is cold or warm, it is impossible to maintain blinding of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold HSG (No Intervention): HSG contrast will be standard, room-temperature
- Warm HSG (Active Comparator): HSG constrast will be warmed.
  Interventions: Drug: Warmed HSG

INTERVENTIONS:
Drug: Warmed HSG — The intervention is warming the HSG constrast.
  Arms: Warm HSG

SUMMARY:
The hysterosalpingogram (HSG) is the gold standard of assessing fallopian tube patency and involves the placement of a transcervical catheter to allow for instillation of radio-opaque dye into the uterine cavity and fallopian tubes which are then imaged with abdominal x-ray. A common side effect of the instillation of dye is the uterine cramping, which is both uncomfortable for the patient as well as can cause iatrogenic proximal occlusion of the fallopian tubes. Proximal tubal obstruction is often not representative of true tubal obstruction but is rather an artifact of the test. Prior studies measuring the perceived pain and cramping during HSG have been conducted which have shown reduced pain scores and decreased uterine cramping when warmed contrast dye is used. The researchers propose that the use of warmed contrast media during HSG will be correlated with decreased pain scores and fewer cases of proximal tubal occlusion in women with otherwise normal uterine anatomy.

DETAILED DESCRIPTION:
Research materials will include obtaining patient past medical history at time of the patient screening and recruitment, via utilization of Epic to search for demographic factors including age, height, weight, BMI, race/ethnicity, duration of infertility, past medical history, and gynecologic/obstetric history.

Post-procedure images from the HSG/report of the HSG findings will be saved in Epic as per usual standard clinical practice. HSG findings will be transcribed with prior demographics/history into a PHI-safe RedCap. No biospecimens will be collected under this protocol.

Patients undergoing fertility treatment that are recommended to undergo HSG as part of their evaluation will be referred to a dedicated research nurse (RN) for eligibility screening and informed consent.

Once found to be meeting inclusion criteria, the patient will be enrolled and scheduled for HSG as appropriate for their menstrual cycle and clinical care. Typically, patients are scheduled during cycle day 5-10 of their menstrual cycle for best study image quality.

Once scheduled, the patient will be randomized to warmed vs cold (room temperature) HSG. The principal investigator will create a computer-generated randomization table (1:1) using block randomization with randomly varying block size of 4 and 6 without stratification. The research coordinator or treating physician will obtain informed consent.

Study team members will have electronic access to the table of randomization within the secure REDCap randomization module and will assign each patient to a single-blinded treatment group once informed consent is obtained.

HSG will be performed in accordance with clinic policy by a physician or physician assistant trained in the procedure and interpretation of study results. Patients will be asked to complete a post-procedure questionnaire.

All data will be collected by the research nurse and entered into RedCap by a member of the study team in a deidentified coded manner.

A single study visit lasting approximately 1 hour will be conducted. This includes the time to meet with the nurse and sign consents and then have HSG procedure performed.

This study will be blinded in a manner that the research nurse, patient, and provider will not be aware of patient allocation at time of recruitment and enrollment. The patient will be assigned a unique study ID number and the randomization module in REDCap will be used to assign the participant to either the experimental (warm) or control (cold) group.

The patient will remain blinded to the treatment allocation but the research nurse and performing provider will be unblinded to allow for correct choice and use of warm versus cold contrast media. As both the research nurse and provider will touch the HSG contrast media and be able to discern if it is cold or warm, it is impossible to maintain blinding of the research team.

The control group (cold contrast) is the current standard of care and is included in this study as a control to allow for comparison with the experimental (warm contrast) group. All patients will obtain an HSG via the same standardized technique at OURM.

Patients may withdraw from the study at any time without repercussions and will be allowed to undergo HSG with standard of care practices at OURM at their discretion. Withdrawal of participation in the study will not change the course of a patient's fertility evaluation or treatment. If the study were to end prematurely, all patients will maintain scheduled appointments for HSG with standard practice methods (cold contrast dye) to be used as per clinic protocol.

All participant recruitment and data collection activities including consenting, interventions, chart reviews, and data analysis will occur at OU Reproductive Medicine clinic (OURM) and via Epic clinical chart review as needed to obtain study data. Data analysis will be conducted in the OUHSC Department of Biostatistics and Epidemiology using data exported from the HIPAA compliant REDCap database and stored on a secure server.

Patients and their fertility provider will all be informed of their HSG results after completion of the procedure as per clinic protocol as part of their fertility evaluation. Patients will be informed of their HSG results after completion of a post-procedure pain questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18-45 undergoing tubal assessment via HSG.

Exclusion Criteria:

1. History of fibroids
2. History of pelvic inflammatory disease (PID or STD including gonorrhea, chlamydia, or trichomonas)
3. History of surgically diagnosed endometriosis or suspected endometriosis on ultrasound (indicated by visualization of likely endometrioma)
4. History of ectopic pregnancy or 3 or more biochemical pregnancies/pregnancy of unknown location
5. History of tubal or ovarian surgery
6. History of known Mullerian anomaly
7. History of pelvic surgery including appendectomy
8. Allergy to iodine-based contrast media
9. History of prior abnormal fallopian tubes on HSG
10. History of ultrasound with hydrosalpinx (unilateral or bilateral)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females of reproductive age will be included, given the nature of HSG.
Enrollment: 240 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-HSG Pain Questionnaire | Measured 1 hour after HSG procedure
  To compare the patient experience for patients undergoing HSG when warm versus cold contrast media is utilized, patients will complete a post-HSG Questionnaire to indicate their level of pain.

SECONDARY OUTCOMES:
Rate of unilateral and bilateral proximal fallopian tube occlusion | Measured at the time of HSG procedure
  The event proportions of unilateral and bilateral proximal fallopian tube occlusion at the time of HSG procedure will be compared between warms versus cold contrast media groups using chi-square tests or Fisher's exact tests as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: LaTasha Craig, MD, Principal Investigator — University of Oklahoma Health Center
Locations (1):
- University of Oklahoma Health Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No